CLINICAL TRIAL: NCT07223827
Title: Handheld Point of Care Electro-Diagnostic Device
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Sergiu Abramovici, Assistant Professor, Indiana University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 28589
Record Dates: First submitted 2025-10-30; First posted 2025-11-03 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Neurologic Findings
MeSH Terms: conditions — Neurologic Manifestations

STUDY DESIGN:
Masking Description: Principal Investigator will be blinded to participant's neurologic diagnosis at enrollment and during procedure, but will see diagnosis in data analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Treatment Arm (Experimental): Participants will be evaluated using the handheld POC device to compare diagnostic data collected vs. clinical diagnostic data
  Interventions: Diagnostic Test: POC EEG

INTERVENTIONS:
Diagnostic Test: POC EEG — The PI will apply the POC investigational device dry electrodes, as well as SOC SSEP stimulator to the participant and run a standardized diagnostic testing sequence, to cover all 4 limbs, spine, and head. The device connects to a laptop via Bluetooth, and the acquired electrodiagnostic data is visualized on the screen. The PI will analyze the acquired data and determine lateralization, localization, and presumed nature of the lesion or pathology causing the patient's symptoms. The direct contact with the participant should take10-20 minutes. The inferred lateralization, localization, and nature of the presumed lesion, will be then documented, to be compared to the diagnostic insight of using SOC diagnostic methods such as CT, MRI, EEG, SSEP, etc. The participant will receive their regular SOC management and a single, brief evaluation using the POC investigational device.

SUMMARY:
There are currently several products offering POC EEG, intended to be deployed on each patient individually and continuously. The investigators propose studying a different approach by using a migrating POC electrodiagnostic device that is deployed directly by the onsite provider and is actively used, like other POC devices, to acquire real-time diagnostic insight and facilitate immediate medical decision making. This can significantly shorten time to treatment which in several neurological and neurosurgical conditions, and thus, can significantly improve patient outcome.

The investigational POC investigational device is based on a handheld limited electrode array, complemented by various stimulation modalities such as SSEP, VEP and BAEP, and potentially other sensors. For this study, the investigators intend to use readily available industry standard stimulators and only use the proposed POC investigational device to acquire and analyze the data. The POC investigational electrodiagnostic prototype was assembled using OpenBCI8 electronic board and electrodes, based on ADS 129X chip by Texas Instruments, that was shown to provide an adequate low-cost solution for electrodiagnostic data acquisition.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years old or above
* Seen inpatient or in outpatient service at IU Health facilities - Methodist Hospital, and the Neuroscience Center, by a Neurology and/or Neurosurgery consultant as part of their SOC.
* The participant has capacity to sign consent or has an assigned LAR (Legally Authorized Representative - Spouse, parent, sibling, etc.) able to consent on their behalf.

Exclusion Criteria:

* Pregnant woman
* PI unblinded by participant or LAR regarding indication or clinical data
* Burns or extensive skin lesions
* Implanted stimulation devices (any)
* Participant without standard imaging and, or other paraclinical SOC investigations to be comparable to the POC investigational device acquired data.
* Significant acute or chronic medical, neurologic, or other illness in the patient that, in the judgment of the PI, could compromise subject safety, limit the ability to complete the study, and/or compromise the objectives of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-01-10 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Outcome 1 | Day 0
  The diagnostic insights acquired using the POC investigation device regarding lateralization (left/right), localization (cerebral - frontal, temporal, parieto-occipital; spinal - cervical, thoracal, lumbosacral; or radicular), and presumed nature of lesion (i.e. ischemia, hemorrhage, space-occupying lesion), are significantly comparable to, and congruent with, the SOC diagnostic insight regarding same parameters (lateralization, localization and presumed etiology) acquired using SOC techniques such as MRI, 10-20 (standard ubiquity used electrode montage) EEG systems, SSEP, etc. The PI will be the only POC investigational device operator, and will be blinded to patient examination, symptoms and SOC investigation results. The PI will be blinded to all EMR data. The investigator then plans to compare the clinical insight obtained by using the POC investigational device, to SOC.
Outcome 2 | Day 0
  The diagnostic insights acquired using the POC investigation device regarding localization (cerebral - frontal, temporal, parieto-occipital; spinal - cervical, thoracal, lumbosacral; or radicular),are significantly comparable to, and congruent with, the SOC diagnostic insight regarding same parameters (lateralization, localization and presumed etiology) acquired using SOC techniques such as MRI, 10-20 (standard ubiquity used electrode montage) EEG systems, SSEP, etc.
Outcome 3 | Day 0
  The diagnostic insights acquired using the POC investigation device regarding the presumed nature of lesion (i.e. ischemia, hemorrhage, space-occupying lesion), are significantly comparable to, and congruent with, the SOC diagnostic insight regarding same parameters (lateralization, localization and presumed etiology) acquired using SOC techniques such as MRI, 10-20 (standard ubiquity used electrode montage) EEG systems, SSEP, etc.

CONTACTS AND LOCATIONS:
Overall Officials: Sergiu Abramovici, MD, Principal Investigator — Indiana University
Locations (1):
- Indiana University Health, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No